CLINICAL TRIAL: NCT00311519
Title: A Phase IIIB Double Blind, Randomized, Placebo-Controlled, Dose-Comparison Study of Subcutaneous Hydration With and Without Human Recombinant Hyaluronidase (HYLENEX) in Volunteer Subjects
Brief Title: A Phase IIIB Dose Comparison Study of Subcutaneous Hydration With and Without Human Recombinant Hyaluronidase (HYLENEX) in Volunteer Subjects
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HZ2-05-04
Record Dates: First submitted 2006-04-04; First posted 2006-04-06 (Estimated); Last update posted 2006-04-06 (Estimated); Status verified 2006-04

CONDITIONS: Healthy
Keywords: Subcutaneous hydration; Hylenex; Hyaluronidase

INTERVENTIONS:
Drug: Hylenex

SUMMARY:
The purpose of this research study to test the effectiveness of a study medication to increase how fast a solution called lactated Ringer's is absorbed when put under the skin subcutaneously. The medication to be studied is an enzyme called hyaluronidase, and is a human recombinant form of the enzyme. The drug company name for this medication is Hylenex. Hylenex was currently an investigational medication at the initiation of the study, but received FDA approval during the study. An investigational medication is a medication or formulation of a medication that is not approved by the United States Food and Drug Administration for use in this country but may be used in studies such as this one.

DETAILED DESCRIPTION:
The study will be conducted in two sequential stages:

Stage 1: Preliminary assessment of mean flow rate and its inter-subject variability, and a comparison to IV infusion. Each subject will receive a SC infusion of 400 mL (from a 0.5 L bag) of Ringer's lactate solution in each upper arm, followed by one IV infusion of 400 mL of Ringer's lactate solution (from a 0.5 L bag). The SC injection sites will be randomized in a double-blinded fashion to receive either 150 units Hylenex or an equal volume of saline placebo injected into a Y-port in the tubing just above the catheter immediately prior to infusion. 24-gauge angiocatheters will be placed symmetrically in the SC space in both proximal upper extremities at the lateral aspect, midline halfway between the olecranon process and the inferoposterior aspect of the acromion, introduced at a 30-degree angle. A 24-gauge angiocatheter will also be placed in a vein in either the left or right forearm (per randomization). In each upper arm, Ringer's lactate solution will be infused SC by gravity (wide open) by placing the top of the fluid in a 0.5 liter bag at a height of 100 cm above the respective angiocatheter sites. After completion of both SC infusions, Ringer's lactate solution will be infused IV by gravity (wide open) by placing the top of the fluid in a 0.5 liter bag at a height of 100 cm above the angiocatheter sites. The flow rate observations in Stage 1 will be used to either confirm or adjust the proposed sample size for Stage 2, if such adjustment is necessary.

Stage 2: Dose-comparison assessment of rate of flow over the range of 150 to 1,500 units of Hylenex. Each subject will receive a SC infusion of 400 mL (from a 0.5 L bag) of Ringer's lactate solution in each upper arm. The SC injection sites will be randomized in a double-blinded fashion to either Hylenex or an equal volume of saline solution injected into a Y-port in the tubing just above the catheter immediately prior to infusion. 24-gauge angiocatheters will be placed symmetrically in the SC space in both proximal upper extremities at the lateral aspect, midline halfway between the olecranon process and the inferoposterior aspect of the acromion, introduced at a 30-degree angle. In each arm, Ringer's lactate solution will be infused SC by gravity (wide open) by placing the top of the fluid in a 0.5 liter bag at a height of 100 cm above the respective catheter sites. Subjects will be dosed in either two or three sequential cohorts.

Cohort 3, at 750 U, to be conducted ONLY if flow rate for Cohort 2 is at least 20% faster than for Cohort 1 without unacceptable toxicity in Cohort 1, or unacceptable toxicity observed in Cohort 2 and not Cohort

In each stage, safety and tolerability will be assessed through physical examination targeted at infusion sites and volume status assessment, vital signs, and adverse events.

Study Medications Hylenex recombinant (hyaluronidase human injection); rHuPH20 (Hylenex is a registered trademark of Baxter International, Inc. or its subsidiaries)

Duration: In both stages of the study, subjects who are successfully screened for the study will receive a single, one-day session of study drug administration followed by parenteral infusions, and then undergo follow-up evaluations at 1 day (in clinic) and 28 days (by telephone) after treatment.

Subject Population: Normal volunteers satisfying all entry criteria.

Planned Total Sample Size: Considering both stages, no more than a total of 70 subjects may be enrolled in this study.

Stage 1: Five evaluable subjects will be enrolled. It is anticipated that no more than a total of 10 subjects will need to be enrolled to provide 5 evaluable subjects. An evaluable subject is one who completes all 3 parenteral infusions. Subjects not meeting this criterion, including those withdrawn prematurely for reasons other than toxicity, will be replaced.

Stage 2: 15 evaluable subjects per cohort will be enrolled. An evaluable subject is one who has completed both SC infusions and has completed protocol-specified assessments sufficient for determination of safety and tolerability. Subjects not meeting these criteria, including those withdrawn prematurely for reasons other than toxicity, will be replaced. Enrollment of Cohort 3 is dependent on findings in Cohorts 1 and 2. Allowing for some non-evaluable subjects in up to three cohorts, each including 15 evaluable subjects, a total of up to 60 subjects may be entered in this Stage 2.

Stopping Rules: Safety monitoring of enrolled subjects will be ongoing and continuous. If signs or symptoms of unacceptable fluid overload occur, the subject will be withdrawn.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females aged 18 to 60 years, inclusive
2. Agreement that there will be no fluid intake for 12 hours prior to the start of the study infusion (except sips of water to take necessary medications)
3. Vital signs (BP, HR, RR) within normal range
4. Metabolic panel (e.g., sodium, potassium, chloride, bicarbonate, BUN, creatinine, glucose, calcium, AST, ALT, alkaline phosphatase, total bilirubin, albumin, and total protein) within normal range within 7 days of infusion
5. Adequate venous access in at least one forearm
6. A negative pregnancy test (if female of child-bearing potential) within 7 days of infusion
7. Decision-making capacity
8. Signed, written IRB-approved informed consent

Exclusion Criteria:

1. Extremity edema
2. Upper extremity pathology that could interfere with study outcome (e.g., cellulitis, lymphatic disorder or prior surgery, pre-existing pain syndrome, previous mastectomy and/or axillary lymph node dissection, etc.)
3. History of cardiovascular disease
4. Rales on lung auscultation
5. Known allergy to hyaluronidase or any other ingredient in the formulation of HYLENEX
6. Known allergy to bee or vespid venom
7. Known coagulopathy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50
Dates: Start 2005-11; Study Completion 2006-01

PRIMARY OUTCOMES:
Average infusion flow rate (mL/hr) derived from the time to infuse 400 mL of lactated ringers

SECONDARY OUTCOMES:
Average SC infusion rate of flow (mL/hr) derived from time required to drain 400 mL from the 500 mL infusate bag, fluid and tubing AND for the arm circumference to return to baseline
Flow rate determined by weight of infusate bag, fluid and tubing at specified timepoints
For SC infusions, change in arm circumference in three locations in the vicinity of the site of infusion
For SC infusions, time from the beginning of infusion until arm circumference returns to baseline
Subject assessment of local discomfort by placing a mark on a 0 100 mm visual analogue scale (VAS) anchored by no discomfort and worst possible discomfort
Local edema assessed by the Investigator on a 0-4 scale
Leakage of fluid at angiocatheter site assessed by the Investigator on a 0-4 scale, prior to infusion, at mid-infusion, at end of infusion, and (for SC infusions), when arm circumference returns to baseline
Subject's global rank-ordered preference for infusion
Investigator's global rank-ordered preference for infusion
Photographic images of the SC infusion sites
Safety and tolerability, based on adverse events and PE including vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Javier T Quesada, OD, Principal Investigator — West Coast Clinical Trials
Locations (1):
- West Coast Clinical Trials, Long Beach, California, United States

REFERENCES:
- [Derived] Thomas JR, Yocum RC, Haller MF, Flament J. The INFUSE-Morphine IIB study: use of recombinant human hyaluronidase (rHuPH20) to enhance the absorption of subcutaneous morphine in healthy volunteers. J Pain Symptom Manage. 2009 Nov;38(5):673-82. doi: 10.1016/j.jpainsymman.2009.03.010. Epub 2009 Oct 12. PMID 19819667